CLINICAL TRIAL: NCT01942603
Title: Minitub: Prospective Registry of Sentinel Node (SN) Positive Melanoma Patients With Minimal SN Tumor Burden Who Undergo Completion Lymph Node Dissection (CLND) or Nodal Observation
Brief Title: Minimal SN Tumor Burden
Acronym: Minitub
Status: Active, not recruiting | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1208-MG
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cutaneous Melanoma
Keywords: Minimal (SN) tumor burden; Stage III; Patients; Lymphnode Dissections
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Observation
- Complete Lymfnode Dissection

SUMMARY:
The purpose of this registry is to collect data in order to discover whether melanoma patients with minimal SN tumor burden should undergo a complete lymph node dissection (CLND) or not.

Currently, if a patient has a positive (or metastatic) SN, this patient will be offered a CLND, which is a surgical intervention aiming to remove all lymph nodes from the same nodal basin as the SN. However, if the positive (or metastatic) SN is only minimally involved, some centers and/or countries do not offer a CLND routinely. As a matter of fact, the CLND procedure does not increase survival for patients with a minimal SN tumor burden, but can add prognostic information, potentially useful in the subsequent decision-making process. However, this is a surgical operation for the patient, which might be accompanied by significant side effects. Moreover, only approximately 20% of patients with a metastatic SN have further lymph node metastases in the same basin, which means that about 4 patients out of 5 will not benefit from a CLND. Thus, there is an urgent need to identify which SN positive patients could be safely spared from a CLND. It has been demonstrated that breast cancer patients with minimal SN tumor burden can be safely managed with nodal observation only, without performing a CLND. There is evidence that the same situation exists in melanoma as well, but this needs to be validated and this is why we are conducting this registry.

The results of this registry will be crucial to establish an accepted standard of care (CLND or nodal observation) for melanoma patients with minimal SN tumor burden.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histological evidence of primary cutaneous melanoma
* Metastases solely confined within the SN:
* in the sub-capsular space (with no parenchymal infiltration) and with a maximum diameter of the largest metastasis not greater than 0.4 mm or
* regardless of the site, any sub-micrometastasis with a maximum diameter not greater than 0.1 mm If there is more than 1 metastatic SN, the patient will be still eligible provided that all involved SN have minimal tumor burden, regardless of the amount of positive SNs and the interested basin

Exclusion Criteria:

* No history of any other malignancy within the past 5 years, except for non-melanoma skin cancer (Basal Cell Carcinomas or Squamous Cell Carcinomas) and in situ cervical cancer
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with minimal SN tumor burden
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2009-07; Primary Completion 2023-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Distant Metastasis Free Interval (DMFI) | 5 years after last patient in

SECONDARY OUTCOMES:
Regional Control Rate (secondary endpoint): | 5 years after last patient in
Relapse Free Interval (RFI) | 5 years after last patient in
Melanoma Specific Survival (MSS) | 5 years after last patient in
Overall Survival (OS) | 5 years after last patient in
Morbidity: rates of wound infections, lymphedema and neurological damage | 5 years after last patient in

CONTACTS AND LOCATIONS:
Locations (22):
- U.Z. Leuven - Campus Gasthuisberg, Leuven, Belgium
- France (3):
  - CHRU de Lille, Lille
  - CHU de Nice - Hopital De L'Archet, Nice
  - Institut Gustave Roussy, Paris
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Universitaetsklinikum - Essen, Essen
  - UniversitaetsMedizin Mannheim, Mannheim
- Italy (3):
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS - Ospedale Busonera, Padua
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Erasmus MC Cancer Institute - location Daniel den Hoed, Rotterdam
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- The Institute Of Oncology, Ljubljana, Slovenia
- Hospital Clinic Universitari, Barcelona, Spain
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (6):
  - Royal Bournemouth Hospital, Bournemouth
  - Cambridge University Hospital NHS - Addenbrookes Hospital, Cambridge
  - Guy's and St Thomas' NHS - St Thomas Hospital, London
  - St George's Hospital NHS Trust, London
  - Norfolk And Norwich Hospital, Norwich
  - St Helens & Knowsley NHS Trust - Whiston Hospital, Prescott